CLINICAL TRIAL: NCT04285632
Title: Efficacy of a Physiotherapy Intervention by Means of Plyometric Exercises in the Improvement of the Dorsal Ankle Flexion and the Strength of the Sural Triceps in the Jump in Basketball Players. A Randomized Clinical Study.
Brief Title: Plyometric Exercises in Ankle Range of Motion and Sural Triceps Strength in the Jump in Basketball Players
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Lockdown
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PLIO
Record Dates: First submitted 2020-02-25; First posted 2020-02-26 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Basketball
Keywords: Basketball; Plyometric Exercise; Range of motion; Randomized clinical trial; Strength Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Each session will last 15 minutes, taking place for 2 days a week, over a period of 4 weeks. The intervention will take place at the beginning of each training session.
  Prior to training, the Counter Movement Jump and Drop Jump exercises will be performed
  Interventions: Other: Plyometrics exercises
- Control group (No Intervention): Athletes included in the control group will continue with their usual warm-up routine.

INTERVENTIONS:
Other: Plyometrics exercises — Counter Movement Jump exercise. The subject will be placed in an upright standing position, with his hands on his hip. It will perform a rapid downward movement in which it will flex the hips and knees and, immediately, a rapid extension of the legs that will result in the maximum vertical jump. During the flight phase the subject will keep the legs straight. The landing will be done with both feet at the same time. The intervention will be carried out for 300 seconds, in 2 series of 30 jumps each and with 3 minutes of rest between series.
  Drop Jump exercise. The players will be placed on a step, standing and with their feet shoulder-width apart. They will drop forward, landing with both feet at the same time. Upon touching the ground they will perform a maximum vertical jump. The intervention will be carried out for 600 seconds, in 2 series of 25 jumps each, and with 3 minutes of rest between series.
  Arms: Experimental group

SUMMARY:
The objective of plyometric exercises is to improve the range of mobility of the ankle, as well as decrease the stiffness of this joint and increase the strength in the sural triceps, by improving the explosive elastic force.

The objective of the study is to assess the efficacy of plyometric exercises in increasing ankle mobility and increasing strength in the sural triceps, in professional female basketball players aged 18 to 40 years.

Randomized, simple blind clinical study. 48 basketball players will be randomized to the two study groups: experimental (they will perform the Counter Movement Jump (CMJ) and Drop Jump (DJ) exercises) and control (they will follow their usual routine). The intervention will last 4 weeks, with 2 weekly sessions of 15 minutes each. The study variables will be: range of dorsal flexion movement of the ankle (goniometry) and strength of the sural triceps (My Jump 2). A descriptive statistical analysis will be performed calculating the main statistical characteristics. The sample distribution will be analyzed with the Kolmogorov-Smirnov test. The changes after each evaluation will be analyzed with the t-student test for related samples and with the ANOVA test of repeated measures the intra and intersubject effect will be observed. Cohen's formula will be used to calculate the effect size.

It is intended to observe improvement in the range of dorsal ankle flexion movement and strength in the sural triceps.

ELIGIBILITY:
Inclusion Criteria:

* Basketball players
* Female
* Federated and professional
* With an age range of 18 to 40 years
* With more than 4 years of basketball sports

Exclusion Criteria:

* Athletes who have been injured in the last two months
* Who suffer an injury during the intervention process
* Have not signed the informed consent document

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline range of motion in ankle dorsal flexion after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  An assessment will be made with a universal goniometer. The evaluation will be carried out according to the protocol indicated by Lang et al. The subject will be placed supine on the stretcher with the knee extended and the foot in a neutral position. The goniometer axis will be placed in the external maleolus, with the goniometer fixed arm following the fibula line, and the mobile arm following the direction of the fifth metatarsal. The unit of measure of this measuring instrument is the degree. A greater number of degrees indicates a greater dorsiflexion of the ankle.

SECONDARY OUTCOMES:
Change from baseline sural triceps strength after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be carried out using the My Jump 2 application. With this test, the height of the jump and its strength will be measured. The subject will be placed in standing position, in front of the evaluator and the camera of the device by placing their hands on the hip. From the static standing position, perform the vertical jump and during the flight phase the subject will keep the legs stretched. The landing will be done with both feet at the same time. The unit of measure of this measuring instrument is the centimeter. A larger number of centimeters indicates greater strength of the lower limb.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain